CLINICAL TRIAL: NCT04574739
Title: Fetal Monitoring by Transabdominal Electrocardiogram Recording: the ELAINE Pilot Project (ELectronic fetAl monitorINg System)
Brief Title: Fetal Monitoring by Transabdominal Electrocardiogram Recording
Acronym: ELAINE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: CSEM Centre Suisse d'Electronique et de Microtechnique SA - Recherche et Developpement (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-01899
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: To Demonstrate That a New Sensor System Can Register Fetal ECG and Distinguish it From Maternal ECG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fetal monitoring by transabdominal electrocardiogram recording

DETAILED DESCRIPTION:
Cardiotocography (CTG), or electronic fetal monitoring (EFM), is the most common procedure used for fetal assessment before and during labour and largely replaced the use of intermittent heart rate auscultation with the Pinard stethoscope or intrapartal analysis of fetal pH by scalp sampling. It relies on acoustic methods in the audible (auscultation) and inaudible range of the sound spectrum (ultrasound). Ever since its introduction in the late 1960s, the benefit of the method has been controversial. Not only the great inter- and intra-observer variability due to visual interpretation of CTG traces seems to be an issue, but also the technical difficulties of the method: data assessment in adipose patients, active fetuses or multiple gestation, confusions between fetal and maternal pulse, assessment during water delivery, strong contractions or changing labour positions of the parturient. It is common knowledge that CTG leads to unnecessary medical interventions such as caesarean section and vaginal-operative deliveries, with the associated health consequences and economic costs.

Despite the continuous progress made in CTG technology in the past 50 years, CTG devices still have drawbacks, namely their bulkiness (including cables and bedside computers), combined with the limited informative value and suboptimal reliability of the measured signals. The assessment can be uncomfortable for the pregnant patient, due to the fact that the patient is bound to a machine and implicitly to the bed, particularly when a longer surveillance is needed. Long periods of immobility can lead to further medical and psychical problems during pregnancy.

Wireless methods of fetal monitoring exist; nevertheless, the technical difficulties of the assessment seem to be more pronounced when these are employed.

Routine continuous monitoring of physiological signals in normal and extraordinary environments provides useful insides for better understanding and modelling of human physiology. Under contract by the European Space Agency (ESA), the Swiss Centre for Electronics and Microtechnology (CSEM) has designed and developed the LTMS system (Long Term Medical System) system. In 2003, ESA commissioned CSEM to do a definition study for a prototype of LTMS. Following the outcomes of this study, in 2006 CSEM built a first prototype (LTMS-2) for ESA, which was validated at Bern University Hospital in 2008. In the subsequent phase (LTMS-3, 2009-2010), CSEM manufactured a set of upgraded systems which were validated in Antarctica (Concordia Station) in 2010 and during the Rio-Tinto field test of the Austrian Space Forum spacesuit simulator in 2011. In 2015, CSEM delivered to ESA a new sensor system (LTMS-S) with yet improved measuring functionalities and higher overall integration in an easy to-wear vest. The system has been shipped to the Concordia Station in Antarctica for the scientific investigation for monitoring the physiological adaptation of manned crews in remote, isolated, and extreme environments. An in-depth clinical validation study at the University Hospital in Lausanne has shown that the performance of the system was within the contractual specifications and that it fulfilled the requirements set by international medical standards.

Although it has initially been proposed to adapt and use LTMS-S for fetal ECG (fECG) measurements, reconsidering the required noise level and resolution to capture fECG, it has been decided to modify and use the ECGi-CDWe system, which has evolved from LTMS-S and belongs to the cooperative sensors family of CSEM. This system outperforms LTMS-S in terms of noise level, resolution, and also number of electrodes that can be connected (>200). The said system has been designed in the frame of an industrial mandate by respecting the requirements of medical device development. Therefore a reduced version of ECGi-CDWe has been developed, hereafter called ELAINE system.

The objective of the proposed project ELAINE is to build a state of the art fetal surveillance system using this technology and by applying electrocardiography (ECG) as main surveillance method. The project leaders believe that this could substantially improve the quality of continuous fetal monitoring before and during labour, in particular in terms of specificity. From measuring a full ECG with the detachable ELAINE sensors instead of heart rate-based CTG, the project leaders expect a higher reliability in the monitoring of the health status of the unborn. The systems based on LTMS technology are unobtrusive and do not require cabling to bedside devices, increasing the maternal comfort.

As mentioned before, the goal of the study is to adapt the ECGi-CDWe technology for fetal surveillance. The full currently existing adult oriented LTMS-S system consists of a Master unit connected to 8 measurement units via 2 cables. Reference and Guard electrode connections are an integral part of the Master unit. The system is powered by a single battery attached to the Master unit. 8 measurement units are powered from the Master unit via the 2 cables connecting them to the Master unit. ELAINE system, being a part of the cooperative sensors family of CSEM, benefits from a simple cabling scheme as opposed to the star topology connection employed in almost any multi-lead ECG measurement systems in the market.

On one hand, the ELAINE sensors are small, unobtrusive and comfortable to wear. On the other hand, they deliver a wide range of detailed signals with high accuracy. The ECG measured with ELAINE contains for example all the information necessary to diagnose arrhythmic heart diseases. The demonstrated high accuracy of the technology will enable the responsible team at CSEM and the project leaders to record full fetal ECGs (fECGs), thus giving a more accurate image of the cardiac health status of the fetus and making interventions more effective. To make diagnoses even more accurate, the sensors developped by CSEM measure a wealth of additional, signals, e.g. body sounds (potential for fetal heart auscultation), muscular activity (ideal for measuring contractions), vibrations (physical activity of the fetus). Finally, the ELAINE technology allows connecting many sensors in a very simple manner (employing only a single two-wire bus for all sensors), making it very easy to simultaneously record signals on different spots of the mother's body.

The ECG monitoring sensors will be tested at the Maternity Ward of the University Hospital of Bern, in a first phase before labour.

A two-step validation has been planned to validate the measurements performed by the ELAINE system: first it will be validated against the non-invasive gold standard to measure fetal heart rate, i.e. CTG, and secondly it will be validated against a conventional ECG system to measure maternal ECG. This two-step validation is justified as follows: CTG can extract fetal heart rate information; however, not the complete ECG morphology. With ELAINE, the project leaders claim to acquire fetal ECG signal rather than only fetal heart rate information. Therefore, a validation only involving CTG will be a partial one. In order to complete the validation, considering that the primary function of the ELAINE system is to acquire ECG signals, it will be validated against a conventional ECG system which acquires maternal ECG. In order to mitigate the risk of perturbation due to simultaneous connection of two ECG systems, measurements will be conducted one after another - with the justification that ECG morphology of a certain individual does not change in the time frame the experiments were conducted. After the registration, the computer will filter and separate the two ECG curves (fetal and maternal), based on the maternal ECG, which is available from the conventional measurement, and on the fetal heart frequency, which is available after registration with CTG.

Validation procedure:

During the first and last quarter of the recording duration, both ELAINE and a conventional CTG system will be connected to the maternal abdomen. Fetal heart rate information acquired by CTG will be compared with the one to be extracted from ELAINE. During the second and third quarters of the recordings, only the ELAINE device will be placed on the maternal abdomen to perform measurements in the absence of the CTG system.

Two measurement electrodes of ELAINE will be connected to the maternal chest. An ECG recording will be performed for 5 minutes. Then a conventional 2-lead ECG will be connected to the maternal chest upon removal of the ELAINE system. An ECG recording of same duration will be performed.

The project leaders believe that the technology developed for ESA in the LTMS series has the potential to fundamentally change EFM, with the end goal to improve the clinical outcomes of deliveries. For this, the project leaders envisage a product which produces more accurate data on the fetal health status than current CTG devices and which is more comfortable to wear. Following the reasoning above, the project leaders think that this can be achieved with ECG measurements. In ELAINE, the project leaders will for the first time demonstrate that the ELAINE technology is appropriate for monitoring fetal health.

ELIGIBILITY:
Inclusion Criteria:

* Physiological pregnancy (no diagnosed fetal malformations or other pathological conditions)
* Physiological CTG registration
* Physiological fetal growth
* No diagnosed cardiac pathology of the mother
* Written informed consent

Exclusion Criteria:

* Start of labour
* Multiple pregnancy
* Pregnancy < 37 weeks of gestation
* Subjects with skin problems in the abdominal area (such as flesh wounds, cuts in the skin, skin rashes, etc.)
* Subjects with implanted electronic devices (pacemaker, defibrillator, etc.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Ten singleton pregnancies with an age of gestation ≥ 37 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
The main objective of our study is to demonstrate that ELAINE sensors can register fetal ECG and distinguish it from maternal ECG, respectively to adapt them (in the CSEM laboratory) for this purpose. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Surbek, Principal Investigator — Frauenklinik Inselspital
Locations (1):
- Frauenklinik Inselspital, Bern, Switzerland